CLINICAL TRIAL: NCT01501812
Title: Evaluation of Generalization Paradigm Patterns Among Different Psychiatric Disorders (Schizophrenia, Affective Spectrum and Anxiety Disorders) - an Open, Single Center, Longitudinal Study
Brief Title: Evaluation of Generalization Paradigm Patterns Among Different Psychiatric Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Other Study IDs: SHA-04-11
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: MDD; Bipolar Disorder; Schizophrenia Disorder; Anxiety Disorder (Panic Disorder or GAD); PTSD
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Anxiety Disorders; Panic Disorder; Generalized Anxiety Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Schizophrenia: Subjects who are suffering from Schizophrenia or Schizoaffective disorder acording to the DSM-IV-R criteria
  Interventions: Behavioral: Generalization pattern
- Control: Healthy subjects without any mental ilness in axis I or II.
  Interventions: Behavioral: Generalization pattern
- Bipolar: Subjects who are suffering from bipolar I or 2 disorder acording to the DSM-IV-R criteria
  Interventions: Behavioral: Generalization pattern
- MDD: Subjects who are suffering from Major Depressive disorder acording to the DSM-IV-R criteria
  Interventions: Behavioral: Generalization pattern
- Anxiety: Subjects who are suffering from Panic disorder or from Generalized Anxiety disorder acording to the DSM-IV-R criteria
  Interventions: Behavioral: Generalization pattern
- PTSD: Subjects who are suffering from Post Traumatic Stress Disorder acording to the DSM-IV-R criteria
  Interventions: Behavioral: Generalization pattern

INTERVENTIONS:
Behavioral: Generalization pattern — During evaluation a conditioning of a tone (conditioning stimulus) and aversive sound ("metal scratch") will conduct (another tone which will be un-conditioning stimulus for control). Generalization patterns will be evaluated, by measuring the differentiation capability between different tones ("neutral" and "aversive") before and after the conditioning, and after extinction phase. The generalization will also be measured by the "generalization curve" that plotted from displaying tones, different from the original tones, and asked the subject whether the current tone is original or new

SUMMARY:
Learning includes the ability to generalize to new situations and respond to similar, yet not identical stimuli. In previous work, focused on stimulus generalization in healthy volunteers, tones that were negatively reinforced induce wider generalization curves than tones that were positively reinforced, and these in turn induce wider curves than neutral memory (Schechtman et al, 2010).

The current study aimed to evaluate those patterns in different clinical disorders (including Schizophrenia, Bipolar disorder, MDD, Anxiety disorders (Panic and GAD) and PTSD, and healthy subjects that would be used as a control), with consideration whether those patterns are unique to any specific disorder or state.

The generalization patterns evaluation would conduct twice though enable to compare the stability of those patterns during the course of the illness (i.e during remission compared to acute state).

The basic paradigm based on conditioning of a tone (sound) with unpleasant noise, and extinction of that conditioning afterword. During the 60 minutes of evaluation, the capability to discriminate between the original tone and similar but not identical tones, and the tendency to categorize similar tones as identical to the original tone. A neutral tone without conditioning will be used as reference. The clinical diagnosis will conduct by a senior psychiatrist, and the state would be evaluated using standard questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Men and women 20-65 years of age.
* Primary DSM-IV diagnosis of Schizophrenia, Schizoaffective, Bipolar (1 or 2) , Major depressive Disorder , Generalized anxiety disorder, panic disorder, post traumatic stress disorder based on SCID and confirmed by a senior psychiatrist, Or subjects without axis I or II diagnosis (control group).
* Capable and willing to provide informed consent. In any case when there is doubt about the patients' capacity to sign an informed consent, an independent doctor will assess the patient capacities to make treatment decisions with the clinical tool MacCAT-T.
* Able to adhere to the evaluation schedule.
* Able to read, hear, write and speak Hebrew.
* Has signed a written informed consent to participate in the study.

Exclusion Criteria:

* Patients with acute, unstable, significant, or untreated medical illness besides schizophrenia, anxiety disorder or affective disorder, including alcohol and drug dependence.
* Subjects with significant cognitive impairment including dementia, history of head injury, mental retardation, or any other cause to "organic" cognitive impairment.
* Current suicidal ideation or history of a suicide attempt in the past six month
* Subjects who were under compulsory hospitalization.
* Subjects with any other dominant axis I or II diagnosis mainly anxiety disorders, which might interfere with the evaluation of the above disorders.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with severe mental disorder in axis one (i.e Schizophrenia, Bipolar, MDD, Anxiety disorder including Panic or Generalized Disorders, PTSD)and healthy subjects that will be used as control- Thirty subjects at each of the groups.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Generalization pattern differentiation | 60 minutes
  Compare the generalization curve and the differentiation between positive, negative and neutral valency bias

SECONDARY OUTCOMES:
State or trait differentiation | 4-24 weeks
  to find the stability of the outcome between the two visits, and whether there is correlation with clinical state and the generalization patterns

CONTACTS AND LOCATIONS:
Overall Officials: Shahak Yariv, MD, Principal Investigator — Shalvata Mental Health Center
Locations (1):
- Shalvat Mental Health Center, Hod HaSharon, Israel